CLINICAL TRIAL: NCT05693506
Title: "Impact of Remote Therapeutic Cooking Workshops in the Management of Adult Patients Living With Obesity on Dietary Balance: Randomized Interventional Study in Stepped Wedge Type Clusters"
Brief Title: Impacts of Remote Cooking Workshops on Patients With Obesity (CuisTO)
Acronym: CuisTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier FH Manhes (Other)
Responsible Party: Principal Investigator, Damien GALTIER, care and prevention research coordinator, Centre Hospitalier FH Manhes
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2021-A00214-37
Record Dates: First submitted 2022-12-22; First posted 2023-01-23 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Impact of Cooking Workshops on Obese Adults

STUDY DESIGN:
Intervention Model Description: Stepped Wedge
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group Arm A (No Intervention): Arm A: Usual care in the investigating hospitals + questionnaires on daily eating habits, feeling of self-efficacy, etc.
- Experimental Group Arm B (Experimental): Arm B: Usual care in the investigating hospitals + Classic cooking workshops (number of 6) + questionnaires on daily eating habits, feeling of self-efficacy, etc.
  Interventions: Other: Cooking workshops
- Experimental Group C (Experimental): Arm C: Usual care in the investigating hospitals + Cooking workshops in the form of culinary challenges (number of 6) + questionnaires on daily eating habits, feeling of self-efficacy...
  Interventions: Other: Cooking workshops

INTERVENTIONS:
Other: Cooking workshops — Cooking workshop in classic form, i.e. with recipes imposed by the dietician on the participants, or cooking workshops in the form of culinary challenges, i.e. without imposed recipes but according to the creativity of the participants
  Arms: Experimental Group Arm B; Experimental Group C

SUMMARY:
The implementation of therapeutic cooking workshops during the management of obesity in hospitals is now well accepted and recognized as of potential interest on the nutritional level but also cognitive and social (DESPORT, 2015; DAGONEAU, 2008). The literature shows that adults participating in cooking workshops are satisfied and acquire cooking skills potentially useful for improving their health (WOLFSON, BLEICH, 2015; CARAHER, 1999). REICKS (2014, 2018) and REES (2012) point out, however, the low methodological quality of most of the studies conducted and, in fact, the effectiveness of therapeutic cooking workshops has not been formally demonstrated by rigorous randomized studies.

The Care and Prevention Research Unit (CRESP) of the Manhès Hospital Center then built a multicenter research protocol to demonstrate the impact of cooking workshops in the care of patients with obesity. The protocol involves 6 hospitals: Georges Pompidou European Hospital (HEGP) University Hospital Center (department of Prof S. CZERNICHOW), PITIE SALPETRIERE University Hospital Center (department of Prof J.M. OPPERT), Cognacq Jay Hospital Center, Forcilles Hospital Center, Bligny Hospital Center and Manhes Hospital Center .

The CuisTO protocol was selected by the PHRIP Jury of the DGOS (General Direction of the Care Offer French Ministry of Health) in 2019 as a high priority project.

The main objective of this research is to evaluate the effectiveness of remote cooking workshops in the management of obesity, through two methods of setting up therapeutic cooking workshops (so-called "classic" workshops and workshops in the form of "culinary challenges") to improve dietary balance in the context of the care of adult patients living with obesity. Dietary balance will be estimated by compliance with the recommendations of the latest National Health Nutrition Program (PNNS-4 2019-2023), "judged" by the PNNS-GS2 score, the consumption of fruits and vegetables, the frequency of cooking and a reduction in the consumption of ultra-processed dishes that have already been prepared.

This is a multicentre, open-label, controlled, comparative intervention study with sequential randomization in clusters (clusters) of the "stepped wedge" type

ELIGIBILITY:
Inclusion Criteria:

* adult able to cook at home,
* BMI greater than or equal to 30 kg/m²,
* Being affiliated or beneficiaries of a social security scheme,
* can be followed on an outpatient basis,
* with physical and mental autonomy to cook,
* having a kitchen in their place of accommodation (home, household, etc.),
* ability to understand French,
* agreeing to answer the various questionnaires,
* having signed the information and consent form
* Patient having the necessary tools for a workshop by videoconference (smartphone, tablet or computer)
* Patient with sufficient connectivity for a videoconference in their kitchen (wifi, 4G network etc.)

Exclusion Criteria:

* patient undergoing bariatric surgery
* patient planning to undergo bariatric surgery within 6 months
* patient who is not affiliated or beneficiary of a social security scheme,
* patient taking part in another experimental research that may interfere with his physical or mental state to cook for the duration of the study.
* patient having treatments that could have an impact on the study criteria will be excluded (treatment with cortisone, neuroleptics, etc.) according to the judgment of the doctors of the departments concerned
* patient with an unstabilized pathology (hyper or hypothyroidism, etc.) that could have an impact on the study criteria according to the judgment of the doctors in the departments concerned
* patient having attended other programs or other cooking workshops (whether therapeutic or not, "chefs' workshop" type) in the last 6 months
* patient having planned to attend other programs or other cooking workshops (whether therapeutic or not, "chefs' workshop" type) apart from those offered during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
daily diet | 3 months
  the daily food balance, consumption of fruits and vegetables, the frequency of cooking and the reduction in the consumption of ultra-processed dishes already prepared.
  These changes will be measured by the PNNS-GS2 score through a dietary survey and a frequency questionnaire (CHALTIEL et al, national health nutrition program
  - guidelines score 2 (PNNS-GS2): development and validation of a diet quality score reflecting the 2017 French dietary guidelines, British Journal of Nutrition, 2019, 122, 331-342)

SECONDARY OUTCOMES:
Self-efficacy | 3 and 6 months
  Increase in the feeling of self-efficacy measured by the SEPOB (Self-Efficacy of the Obese Patient) Obesity-specific Feeling of Self-Efficacy questionnaire (DESCAMPS J et al., 2010) , measures the specific feeling of self-efficacy related to weight management usable in obese, overweight or normal weight subjects
Patient goals | 3 months
  Achievement of the objectives set by the patient when he participates in a series of 6 cooking workshops such as "I would like to learn to cook vegetables" or "cook less fat". The patient completes a questionnaire (before-after) proposing different possible objectives that the patients would like to achieve by participating in a cooking workshop. When filling out the questionnaire, the patient will have to choose the 3 objectives (out of 12 proposed + 1 free) which seem important to him when he attends a cooking workshop. He will have to number from 1 to 3 the order of importance of his objectives and note on a scale of 1 to 10 the skills he thinks he has in this area. The result is given in terms of the percentage of patients who have reached their initial personalized objective(s) after the two stages of the intervention. The achievement of the objectives set will be considered as achieved if the mark between the two interventions has increased.
BMI | 3 and 6 months
  Patient weight and height (Body Mass Index)

CONTACTS AND LOCATIONS:
Overall Officials: Damien GALTIER, Principal Investigator — Centre Hospitalier FH Manhès
Locations (6):
- France (6):
  - CH Bligny, Briis-sous-Forges
  - Hôpital FORCILLES, Férolles-Attilly
  - CH Manhès, Fleury-Mérogis
  - La Pitié Salpêtrière AP-HP.Sorbonne Université, Paris
  - HEGP, Paris
  - Hôpital Cognacq-Jay, Paris

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT05693506/Prot_SAP_000.pdf